CLINICAL TRIAL: NCT03673748
Title: Phase II, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate Safety and Efficacy of Mesenchymal Stem Cells (MSV-allo) in the Treatment of Lupus Nephritis
Brief Title: Treatment of Lupus Nephritis With Allogeneic Mesenchymal Stem Cells
Acronym: MSV_LE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Red de Terapia Celular (Industry)
Collaborators: Hospital del Rio Hortega (Other); Hospital Clínico Universitario de Valladolid (Other); University of Valladolid (Other); Citospin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TerCel_006; 2022-000243-80 (EudraCT Number)
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Lupus Nephritis; Lupus Erythematosus
Keywords: Lupus Erythematosus; Lupus Nephritis; Stem Cell; Mesenchymal Stem Cells; Autoimmune diseases; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Nephritis; Autoimmune Diseases; Lupus Erythematosus, Systemic | interventions — Genes, mos; Saline Solution

STUDY DESIGN:
Intervention Model Description: Control arm (placebo) and experimental arm (mesenchymal stem cells)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both Experimental and Control arms will receive a similar endovenous injection with either cells or placebo. Blind to participant, investigator and care providers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mesenchymal stem cells (MSC) (Experimental): Participants will receive a single Intravenous infusion of Mesenchymal Stem Cells (MSV) 2 million cells per kg wt suspended in 100 ml of physiological saline solution. All participants will receive the infusion at the Baseline (Day 0) visit. All participants will continue on their standard-of-care therapy during the trial. GMP-compliant MSV will be prepared by IBGM-University of Valladolid-Citospin.
  Interventions: Drug: Mesenchymal stem cells (MSC)
- Placebo (Placebo Comparator): Participants will receive a placebo infusion (100 ml of physiological saline solution) that does not contain any mesenchymal stem cells.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mesenchymal stem cells (MSC) — Endovenous injection of MSV in saline solution
  Other Names: MSV, GMP-compliant MSC manufactured by IBGM in Valladolid
  Arms: Mesenchymal stem cells (MSC)
Drug: Placebo — Endovenous injection of saline solution without cells
  Other Names: Saline solution
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mesenchymal stem cells (MSCs) obtained from bone marrow for the treatment of adults with active proliferative lupus nephritis. The objective of this study is to evaluate the efficacy of mesenchymal stem cells (MSCs) in achieving a full or partial response in the treatment of Lupus Nephritis (LN) during its induction period.

DETAILED DESCRIPTION:
A Phase 2b, double-blind (neither the participant nor the investigator will know if active drug or placebo is assigned), placebo-controlled, randomized (assigned by chance), in which subjects with Lupus Nephritis (LN), who do not respond -or respond partially- to induction treatment, shall receive either MSCs (2 million cells/Kg) or placebo by intravenous injection. The administration of cells will be done only once.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Females or males ≥18 years old who provide written informed consent at the selection visit.
2. Diagnosis of systemic lupus erythematosus (SLE) by meeting at least 4 of the 11 criteria included in the American College of Rheumatology (ACR) classification and/or the Systemic Lupus International Collaborating Clinics (SLICC) criteria, at the selection visit.
3. Diagnosis of lupus nephritis (LN) using the 2003 classification of the International Society of Nephrology and the Society of Renal Pathology, by biopsy performed no more than 6 months before the selection visit if they enter from the induction period, and no more than one year if they enter with a moderate/severe recurrence.
4. No response or partial response to standard treatment, or moderate/severe recurrence of lupus nephritis.
5. SLEDAI-2K ≥ 10 during the selection period.
6. Women of childbearing potential should use effective methods of contraception to prevent pregnancy.
7. Have been vaccinated against pneumococcus and influenza at the time the vaccination campaign is carried out.

EXCLUSION CRITERIA:

A - Related to previous treatments:

1. Use of corticosteroids or mycophenolate above the doses allowed for induction, according to the Consensus Document of the Systemic Autoimmune Diseases Group of the Spanish Society of Internal Medicine and the Spanish Society of Nephrology.
2. Use of rituximab, belimumab, ocrelizumab or other biologic therapies against B cells in the 6 months prior to selection.
3. Use of cyclophosphamide in the 6 months prior to selection.
4. Use of any tumor necrosis factor inhibitor treatment in the 6 months prior to selection.
5. Use of immunoglobulins in the 6 months prior to selection.
6. Change in doses of an angiotensin converting enzyme inhibitor or an angiotensin receptor inhibitor in the two months prior to selection.
7. Treatment with another investigational medicinal product within three months prior to selection or 5 times the half-life of the agent.

   B - Related to medical problems:
8. Any pathology, including an uncontrolled disease other than SLE, which, in the opinion of the investigator, the sponsor or the person they designate, constitutes an inappropriate risk or a contraindication for participation in the trial or that could interfere with the objectives of the trial, its performance or evaluation.
9. Cardiac, peripheral, or cerebrovascular cardiovascular events in the 6 months prior to the selection visit.
10. Active cardiac arrhythmia or clinically significant electrocardiogram abnormalities at selection visit or on the day of randomization that, in the opinion of the investigator, sponsor, or designee, constitute an inappropriate risk or contraindication to participation in the study.
11. Thromboembolic events in the 12 months prior to or during selection, whether or not associated with associated antiphospholipid syndrome, or inadequate anticoagulation tests 6 weeks immediately prior to or during selection visit.
12. Active central nervous system SLE that is considered severe or progressive (recent uncontrolled seizures, changes in anticonvulsant treatment within 3 months prior to selection visit, or resulting in significant cognitive impairment).
13. History or current diagnosis of a demyelinating disease such as multiple sclerosis or optic neuritis.
14. Comorbidities that require treatment with systemic corticosteroids (oral, rectal or injectable) such as asthma or inflammatory bowel disease.
15. Antecedents or plans for an organ transplant.
16. Clinically significant active viral, bacterial or fungal infection, or having suffered a major episode of infection that required hospitalization or parenteral treatment in the 4 weeks prior to the selection visit, during the selection visit, or having finished anti-infective treatment within 2 weeks prior to or during selection, or a history of recurrent infections (three or more cases of the same type of infection in a consecutive 12-month period). Controlled vaginal candidiasis, onychomycosis, and genital or oral herpes simplex virus would not be reasons for exclusion.
17. History of or positive human immunodeficiency virus (HIV) test result, hepatitis C antibodies and/or detection by polymerase chain reaction, hepatitis B surface antigen (HBsAg+), and/or IgM or total antibodies against hepatitis B nuclear antigen at selection.
18. Diagnosis of active or latent tuberculosis (TB) using a purified protein derivative TB skin test (induration ≥ 5 mm) or a positive Quantiferon test result, at selection or within 3 months prior to the selection visit. Patients who have completed previous adequate treatment or who are receiving treatment will not repeat the test. Patients who are receiving adequate TB treatment for at least 4 continuous weeks prior to the selection visit and who are expected to complete the treatment regimen will not be excluded.
19. Presence of class 3 or 4 uncontrolled congestive heart failure according to the New York Heart Association.
20. Active cancer.
21. Major surgical intervention within 6 weeks prior to selection visit or planned during the trial period, including follow-up.
22. Pregnant or lactating women.

    C - Laboratory abnormalities:
23. Clinically significant laboratory test abnormalities not attributed to active SLE.
24. Chest X-ray with significant changes indicating active TB. The chest X-ray must have been performed within 3 months prior to the selection visit or during the selection period.

    D - Others:
25. Legal incapacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have achieved complete response | 0-24 weeks
  Complete renal response criteria: glomerular filtration rate ≥ 60ml/min/1.73m², or decrease to initial values or ± 15% of the baseline value in those with glomerular filtration rate < 60ml/min/1.73m²; proteinuria ≤ 0.5 g/24h; inactive sediment: ≤ 5 red blood cells, ≤ 5 leukocytes, absence of red blood cell casts; and serum albumin > 3 g/dl.
Proportion of patients who have achieved partial response | 0-24 weeks
  Partial renal response criteria: if baseline proteinuria ≥ 3.5 g/24h, decrease in proteinuria < 3.5 g/24h; if baseline proteinuria < 3.5 g/24h, proteinuria reduced by > 50% compared to baseline; in both situations stabilization (±25%) or improvement in glomerular filtration compared to baseline values.

SECONDARY OUTCOMES:
Proportion of patients at week 24 whose prednisone-equivalent corticosteroid dose has been reduced | 0-24 weeks
  The corticosteroid reduction is defined as reduction by ≥ 25% in comparison with the selection visit and to a dose ≤ 7.5 mg/day and who have no exacerbation BILAG A or 2B. A BILAG A or 2B exacerbation is defined as at least one new BILAG A organic domain score or at least 2 new BILAG B organic domain scores compared to the selection visit.
Proportion of patients at each visit whose prednisone-equivalent corticosteroid dose has been reduced | Throughout the study until its completion, an average of 1.5 years
  The corticosteroid reduction is defined as reduction by ≥ 25% in comparison with the selection visit and at a dose ≤ 7.5 mg/day, and who do not have any BILAG A or 2B exacerbations of disease activity.
Proportion of patients at week 24 with a specific reduction relative to the selection visit in the daily dose of prednisone-equivalent corticosteroids. | 0-24 weeks
  Different levels of corticosteroid dose reduction: 0-<25%, 25%-50%, >50%.
Cumulative dose of corticosteroids | 0-24 weeks
  Cumulative dose of corticosteroids equivalent to prednisone up to week 24
Proportion of patients who have reduced the dose of immunosuppressants | 0-24 weeks
  Proportion of patients who, up to week 24, have reduced the dose of immunosuppressants without presenting any BILAG A or 2B exacerbation.
Change from baseline in SF-36 score | Throughout the study until its completion, an average of 1.5 years
  Quality of life questionnaire (SF-36)
Change from baseline in LupusQoL score | Throughout the study until its completion, an average of 1.5 years
  Quality of life questionnaire specific for LES (LupusQoL)
Change in proteinuria levels | Throughout the study until its completion, an average of 1.5 years
  Change from baseline in the levels of proteinuria, a sign of disease activity
Change in disease activity (SLEDAI-2K index) | Throughout the study until its completion, an average of 1.5 years
  Change in disease activity measured by change from baseline of Systemic Lupus Erythematosus Disease Activity (SLEDAI-2K) index, which computes the score of different parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Barbado, MD, PhD, Study Chair — University Hospital Río Hortega, Valladolid, Spain; Rosa Conde, PhD, Study Director — University Hospital Río Hortega, Valladolid, Spain; Margarita González-Vallinas, PhD, Principal Investigator — University of Valladolid
Locations (1):
- University Hospital Río Hortega, Valladolid, Valladolid, Spain

REFERENCES:
- [Background] Vega A, Martin-Ferrero MA, Del Canto F, Alberca M, Garcia V, Munar A, Orozco L, Soler R, Fuertes JJ, Huguet M, Sanchez A, Garcia-Sancho J. Treatment of Knee Osteoarthritis With Allogeneic Bone Marrow Mesenchymal Stem Cells: A Randomized Controlled Trial. Transplantation. 2015 Aug;99(8):1681-90. doi: 10.1097/TP.0000000000000678. PMID 25822648
- [Background] Noriega DC, Ardura F, Hernandez-Ramajo R, Martin-Ferrero MA, Sanchez-Lite I, Toribio B, Alberca M, Garcia V, Moraleda JM, Sanchez A, Garcia-Sancho J. Intervertebral Disc Repair by Allogeneic Mesenchymal Bone Marrow Cells: A Randomized Controlled Trial. Transplantation. 2017 Aug;101(8):1945-1951. doi: 10.1097/TP.0000000000001484. PMID 27661661
- [Background] Barbado J, Tabera S, Sanchez A, Garcia-Sancho J. Therapeutic potential of allogeneic mesenchymal stromal cells transplantation for lupus nephritis. Lupus. 2018 Nov;27(13):2161-2165. doi: 10.1177/0961203318804922. Epub 2018 Oct 5. PMID 30290717
- See also: SLE — https://ghr.nlm.nih.gov/condition/systemic-lupus-erythematosus
- See also: Lupus — https://medlineplus.gov/lupus.html